CLINICAL TRIAL: NCT00242346
Title: A Double-Blind, Randomised, Dose Ranging, Multi-Centre, Phase IIIb Study to Evaluate the Efficacy and Safety of High Doses of Candesartan Cilexetil (Atacand®) on the Reduction of Proteinuria in the Treatment of Subjects With Hypertension and Moderate to Severe Proteinuria
Brief Title: High Doses of Candesartan Cilexetil on the Reduction of Proteinuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D2452L00006; DC-AHS-0006; SMART
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Proteinuria
Keywords: Hypertension
MeSH Terms: conditions — Proteinuria; Hypertension | interventions — candesartan cilexetil

INTERVENTIONS:
Drug: candesartan cilexetil

SUMMARY:
The purpose of this study is to assess the effects of high doses of candesartan cilexetil and also to assess which dose (16mg, 64mg, 128mg) is the most optimal for the maximum reduction of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Stable hypertension defined as no new antihypertensive medication started within 6 weeks of Visit 1
* Minimum 6-month history of hypertension and primary glomerular disease
* Hypertensive nephrosclerosis
* Diabetic nephropathy with stable proteinuria as defined by ≥ 1g/24 hours on more than one occasion within 6 months prior to Visit 1

Exclusion Criteria:

* Persistent hypertension
* New anti-hypertensive medications started within 6 weeks of Visit 1
* Significant cardiac disease or Liver disease
* Females of childbearing potential without reliable contraception
* Pregnant women and women who are breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2003-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine the effects of high dose candesartan cilexetil on the overall reduction in proteinuria from baseline as evidenced by the 24-hour urine collection

SECONDARY OUTCOMES:
To determine the effects of high dose candesartan cilexetil on renal function as measured by serum creatinine and 24-hour creatinine clearance
To determine the effects of high dose candesartan cilexetil on blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Kazi Borkowski, PhD, Study Director — AstraZeneca; Norman MuirHead, MD, Principal Investigator — London HSC; Ellen Burgess, MD, Principal Investigator — Foothills Medical Center
Locations (26):
- Canada (26):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Courtice, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Richmond Hill, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Timmins, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Weston, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Ste-Foy, Quebec
  - Research Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Cooper TE, Teng C, Tunnicliffe DJ, Cashmore BA, Strippoli GF. Angiotensin-converting enzyme inhibitors and angiotensin receptor blockers for adults with early (stage 1 to 3) non-diabetic chronic kidney disease. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD007751. doi: 10.1002/14651858.CD007751.pub3. PMID 37466151
- [Derived] Burgess E, Muirhead N, Rene de Cotret P, Chiu A, Pichette V, Tobe S; SMART (Supra Maximal Atacand Renal Trial) Investigators. Supramaximal dose of candesartan in proteinuric renal disease. J Am Soc Nephrol. 2009 Apr;20(4):893-900. doi: 10.1681/ASN.2008040416. Epub 2009 Feb 11. PMID 19211712